CLINICAL TRIAL: NCT04800081
Title: Effect of Sacubitril/Valsartan on Urinary Microalbumin and Pulse Wave Velocity in Perimenopausal Patients With Hypertension
Brief Title: Effect of LCZ696 on Urinary Microalbumin and Pulse Wave Velocity in Perimenopausal Patients With Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Ying Pei, house physician, LanZhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020A-247
Record Dates: First submitted 2021-03-01; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Hypertension
Keywords: perimenopausal; hypertensive; Sacubitril/Valsartan; pulse wave velocity; urinary microalbuminuria
MeSH Terms: conditions — Hypertension | interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Intervention Model Description: A total of 264 cases of perimenopausal patients with essential hypertension who were admitted to Department of Cardiology, Second Hospital of Lanzhou University,from January, 2020 to March,2021 will be enrolled and randomized to receive once-daily treatment with 100-400 mg of Sacubitril/Valsartan or 80-320 mg of Valsartan.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sacubitril/Valsartan (Experimental): receive once-daily treatment with 100-400 mg of Sacubitril/Valsartan
  Interventions: Drug: Sacubitril/Valsartan
- Valsartan (Active Comparator): receive once-daily treatment with 80-320 mg of Valsartan
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril/Valsartan — Patients will be randomized to receive once-daily treatment with 100-400 mg of Sacubitril/Valsartan.
  Other Names: LCZ696
  Arms: Sacubitril/Valsartan
Drug: Valsartan — Patients will be randomized to receive once-daily treatment with 80-320 mg of Valsartan.
  Other Names: Diovan
  Arms: Valsartan

SUMMARY:
To explore the efficacy of Sacubitril/Valsartan in the treatment of perimenopausal hypertensive patients, as well as the difference between the antihypertensive efficacy and valsartan, the therapeutic effect of its exposure to different factors and the protection of target organs.To provide reference for the clinical treatment of perimenopausal hypertension patients with shakubactrivalsartan.

1. To evaluate the effects of Sacubitril/Valsartan on urinary microalbumin and pulse wave velocity in perimenopausal hypertension patients.
2. To evaluate the clinical application of Sacubitril/Valsartan in the treatment of perimenopausal hypertension, so as to improve the blood pressure management ability and control rate of patients with such hypertension.

DETAILED DESCRIPTION:
A total of 264 cases of perimenopausal patients with essential hypertension who were admitted to Department of Cardiology, Second Hospital of Lanzhou University,from January, 2020 to March,2021 will be enrolled and randomized to receive once-daily treatment with 100-400 mg of Sacubitril/Valsartan or 80-320 mg of Valsartan.The general information, menstrual history, cardiac ultrasound, urinal-renal function, PWV, baseline blood pressure, post-medication blood pressure, whether to use antihypertensive drugs and the type of antihypertensive drugs of the patients were enrolled.After 12 weeks of drug intervention, left ventricular mass indexwere measured by cardiac ultrasound, PWV, urinary microalbinin, 24-hour ambulatory blood pressure monitoring, biochemical indicators will be collected.SPSS22.0 statistical software was used for statistical analysis of PWV, urinary microalbumin, blood pressure and other results by paired data t-test, and the chi-square test was used for non-count data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with essential hypertension（SBP>140 and <180 mmHg, and/or DBP>90 and <110 mmHg)）were diagnosed according to the hypertension diagnostic criteria of the Chinese Guidelines for Hypertension (2018 Revised Edition)；
2. Female aged 45-55 years old and meeting the perimenopausal criteria in the STRAE+10;
3. No other complications, no treatment or ongoing antihypertensive therapy (SBP ≥140mmHg or Diastolic BP ≥90mmHg)；
4. Agree to participate in the study and sign the informed consent；

Exclusion Criteria:

1. Secondary hypertension；
2. History of angioedema；
3. Heart failure NYHA grade III or above (excluding grade III)；
4. Liver and kidney dysfunction (ALT or AST≥ three times the upper limit of normal value, that is, ALT≥120U/L,AST≥120U/L, creatinine clearance < 30ml/min);
5. Hyperkalemia (serum potassium ≥5.5mmol/L);
6. Moderate or above anemia (HGB≤90g/L);
7. Bilateral renal artery stenosis;
8. History of stroke;

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-06-09 (Estimated); Study Completion 2021-07-09 (Estimated)

PRIMARY OUTCOMES:
Blood pressure，24 hour automatic blood pressure monitoring，home blood pressure monitoring，Office blood pressure | Evaluation at 12 weeks of treatment will be reported
  Changes in this major indicators were detected before and after drug treatment in both groups
urinary microalbuminuria | Evaluation at 12 weeks of treatment will be reported
  Changes in this major indicators were detected before and after drug treatment in both groups
pulse wave velocity | Evaluation at 12 weeks of treatment will be reported
  Changes in this major indicators were detected before and after drug treatment in both groups
ventricular mass indexwere measured by cardiac ultrasound | Evaluation at 12 weeks of treatment will be reported
  Changes in this major indicators were detected before and after drug treatment in both groups

SECONDARY OUTCOMES:
Adverse events | During the drug intervention up to 30 days,60 days and 80days,it will bereported in the final.
  such as arrhythmology，dizzy， headache，edema，cough.Other incidents are even more serious

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Second Hospital of Lanzhou University, Lanzhou, GuSu, China